CLINICAL TRIAL: NCT00514449
Title: A Randomized Double-blind Controlled Trial of Valacyclovir Add-on Treatment of HSV Positive Early Course Schizophrenia Patients
Brief Title: Systematic Evaluation of Antiviral Medication in Schizophrenia
Acronym: SEAMS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Konasale Prasad (Other)
Collaborators: Stanley Medical Research Institute (Other); Wayne State University (Other)
Responsible Party: Sponsor-Investigator, Konasale Prasad, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0602032
Record Dates: First submitted 2007-08-08; First posted 2007-08-10 (Estimated); Results first posted 2018-05-09 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Valacyclovir (Experimental): 1 gram pill taken twice a day for 2 weeks, after 2 weeks it increased to 1.5 gram pill taken twice a day for 16 weeks.
  Interventions: Drug: Valacyclovir
- Sugar pill (Placebo Comparator): 2 placebo pills taken twice a day for 2 weeks, after 2 weeks 3 pills taken twice a day for 16 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valacyclovir — 1 g PO BID x 2 weeks after 2 weeks it goes up to 1.5 g PO BID x 16 weeks along with antipsychotic
  Arms: Valacyclovir
Drug: Placebo — 2 pills twice a day x 2 weeks, after 2 weeks 3 pills twice a day x 16 weeks along with antipsychotic
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to examine whether antiviral medication will help improve psychotic symptoms and cognition in individuals early in the course of schizophrenia or schizoaffective disorder who are exposed to herpes simplex virus, type 1 (HSV 1), a virus that causes commonly occurring and recurrent cold sores.

DETAILED DESCRIPTION:
The main objective of the study is to evaluate the efficacy of add-on treatment of Valacyclovir (VAV), an antiviral medication, in the treatment of early course schizophrenia/schizoaffective disorder patients. Our main hypothesis is that the VAV add-on treatment will improve positive, negative and cognitive symptoms in herpes simplex virus (HSV) positive schizophrenia or schizoaffective disorder patients. We hypothesize that the grey matter reductions in specific brain regions (such as prefrontal regions) will improve in patients on VAV + antipsychotic compared to those on placebo + antipsychotic and the improvements in positive, negative and cognitive symptoms will be correlated with the grey matter changes.

ELIGIBILITY:
Inclusion Criteria:

* Both genders between the ages of 18-50 years
* Schizophrenia or schizoaffective disorder as defined in DSM-IV
* Duration of illness 10 years or less
* On a stable dose of an antipsychotic medication for at least a month
* Should score 4 or more on at least one of the subscales of PANSS
* Positive for HSV1
* Written informed consent

Exclusion Criteria:

* Substance abuse in the last month/dependence 6 months prior to the study
* History of, or current medical/neurological illnesses which affects CNS function e.g., epilepsy, head injury with prolonged loss of consciousness
* Pregnancy
* History of immune disorders, HIV infection or currently receiving immunosuppressants
* Subjects on regular antiviral therapy
* History of hypersensitivity to Valacyclovir
* Mental retardation as defined in DSM-IV

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2007-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Konasale Prasad, MD, Principal Investigator — Western Psychiatric Institute and Clinic; Vishwajit Nimgaonkar, MD, PhD, Principal Investigator — Western Psychiatric Institute and Clinic; Matcheri Keshavan, MD, Principal Investigator — Wayne State University; Rajaprabhakaran Rajarethinam, MD, Principal Investigator — Wayne State University
Locations (2):
- United States (2):
  - Wayne State University, Detroit, Michigan
  - Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Prasad KM, Shirts BH, Yolken RH, Keshavan MS, Nimgaonkar VL. Brain morphological changes associated with exposure to HSV1 in first-episode schizophrenia. Mol Psychiatry. 2007 Jan;12(1):105-13, 1. doi: 10.1038/sj.mp.4001915. Epub 2006 Oct 10. PMID 17033628
- [Derived] Prasad KM, Eack SM, Keshavan MS, Yolken RH, Iyengar S, Nimgaonkar VL. Antiherpes virus-specific treatment and cognition in schizophrenia: a test-of-concept randomized double-blind placebo-controlled trial. Schizophr Bull. 2013 Jul;39(4):857-66. doi: 10.1093/schbul/sbs040. Epub 2012 Mar 23. PMID 22446565

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between 7/2007 and 8/2009 at two separate sites, Pittsburgh and Detroit. Recruitment took place through the local hospital and community mental health and school counseling centers, as well as other research studies and area mental health conferences.
Pre-assignment Details: Patients first had a placebo run-in for two weeks along with the psychiatric medications they were on and then randomized at Week 2 to either VAV or placebo group. Enrolled subjects were excluded due to cannabis abuse, claustrophobia, and a duration of illness that was too long.
Period: Overall Study
Arm/Group | Valacyclovir | Sugar Pill
Started | 12 | 12
Completed | 9 | 8
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Protocol Violation | 1 | 2
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valacyclovir | Sugar Pill | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (9.4) | 28.7 (8.5) | 29.2 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: PANSS Positive and Negative Syndrome Scale for Schizophrenia
Description: This is a structured measure of severity of psychopathology that includes both positive and negative symptoms. The range is a minimum score of 30 and the maximum is 210. The lower scores suggest milder severity of illness domains.
Time Frame: Baseline, Weeks 2, 4, 6, 10, 14, 18
Population: Comparative analysis of active drug versus placebo
Measure: Mean (Standard Deviation); unit: Scores on the scale
Arm/Group | Valacyclovir | Sugar Pill
Number analyzed (Participants) | 12 | 12
Scores on the scale
  Scores at Baseline of the trial | 70.08 (12.616) | 83.92 (13.895)
  Scores at week 2 of the trial | 72.25 (11.450) | 77 (14.917)
  Scores at week 4 of the trial | 67.36 (12.314) | 75.2 (13.998)
  Scores at week 6 of the trial | 65.583 (9.228) | 74.3 (16.275)
  Scores at week 10 of the trial | 65.2 (10.737) | 73.2 (12.044)
  Scores at week 14 of the trial | 57.1 (12.511) | 69.6 (14.886)
  Scores at the end of the trial | 56.5 (9.289) | 67.125 (13.726)

2. Primary Outcome: Cognitive Function Neuropsychological Battery (Gur Battery)
Description: All results are given as the mean difference between an 18 week follow-up and the baseline battery administrations.This is a computerized test that measures both accuracy and response times. A range for response times is not available because of individual variabilities. Accuracy scores can vary for each test: Working memory accuracy range was 0-16. Verbal memory accuracy range was 0-20. For both, the higher the score the better. No cut offs are available
Time Frame: Baseline, Week 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Valacyclovir | Sugar Pill
Number analyzed (Participants) | 12 | 12
units on a scale
  Working Memory: 2-Back Test Accuracy | 2.13 (2.68) | 0.13 (2.9)
  Immediate Verbal Memory Reaction Accuracy | 2.44 (2.62) | -0.49 (3.11)

3. Secondary Outcome: Changes in Grey Matter Deficit
Description: Gray matter volume changes (in cc) were measured using structural MRI. Changes were reported as gray matter volume in cc. Note: Assessment of blood oxygenation level dependent (BOLD) changes using fMRI were erroneously included in the original study record.
Time Frame: Baseline, Week 18
Population: Analysis included on all participants on whom baseline and week 18 data were collected. Valacyclovir and placebo groups
Measure: Mean (Standard Deviation); unit: cm^3
Groups:
- Valacyclovir: A time by treatment group interaction showed increased gray matter volume estimated as number of voxels in a cluster with Valaclcovir compared to placebo
- Sugar Pill: A time by treatment group interaction showed decreased or no significant change in the gray matter volume estimated as number of voxels in a cluster with Valaclcovir compared to placebo
Arm/Group | Valacyclovir | Sugar Pill
Number analyzed (Participants) | 9 | 8
cm^3 | 26.83 (5.04) | 24.22 (2.85)
Statistical Analysis 1: Comparison: Valacyclovir vs Sugar Pill; Test type: Other; p = 0.004, ANCOVA — p value is adjusted for multiple comparisons; number of voxels in a cluster = 2037 — Time by treatment group interaction term

ADVERSE EVENTS:
Time Frame: 2, 4, 6, 10, 14, and 18 weeks.
Arm/Group | Valacyclovir | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 5/12 | 6/12
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valacyclovir (N=12) | Sugar Pill (N=12)
Stomach Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Mild Extrapyramidal Symptoms (Psychiatric disorders) | 0 (0) | 1 (1)
Pain in Elbow when Extended (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Increased Sexual Drive (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Leg Cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Motion Sickness (Nervous system disorders) | 1 (1) | 0 (0)
Tongue Twitch (Nervous system disorders) | 1 (1) | 0 (0)
Slight Tremor (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This was a small sample study designed as a proof of concept. A larger study will follow.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No